CLINICAL TRIAL: NCT02242370
Title: An Open-label Evaluation of the Effectiveness of MICARDIS® (Telmisartan) on Blood Pressure Control and Quality of Life in Patients With Essential Hypertension The MICARDIS COMMUNITY ACCESS TRIAL (MicCAT)
Brief Title: Effectiveness of MICARDIS® (Telmisartan) on Blood Pressure Control and Quality of Live in Patients With Essential Hypertension
Acronym: MicCAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 502.461
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

ARMS (2):
- Telmisartan low dose (Experimental)
  Interventions: Drug: Low dose of telmisartan
- Telmisartan high dose (Experimental)
  Interventions: Drug: High dose of telmisartan

INTERVENTIONS:
Drug: Low dose of telmisartan
  Arms: Telmisartan low dose
Drug: High dose of telmisartan
  Arms: Telmisartan high dose

SUMMARY:
Study to assess the effect of Telmisartan on diastolic and systolic blood pressure and to establish the effect on patient's quality of life scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Stage I essential Hypertension (diastolic blood pressure 90-99 mmHg, and/or systolic blood pressure 140-159 mmHg)
* Signed informed consent form

Exclusion Criteria:

- Females of childbearing potential

Ages: 20 Years to 93 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3045 (Actual)
Dates: Start 1999-09; Primary Completion 2000-11 (Actual)

PRIMARY OUTCOMES:
Change in diastolic blood pressure | Pre-dose, up to 6 weeks after start of treatment
Change in systolic blood pressure | Pre-dose, up to 6 weeks after start of treatment
Changes from baseline in the quality of life (QOL) scores by patient self-assessment | Pre-dose, 6 weeks after start of treatment

SECONDARY OUTCOMES:
Assessment of blood pressure control rate | Up to 6 weeks after start of treatment
Assessment of systolic blood pressure response rate | Up to 6 weeks after start of treatment
Assessment of diastolic blood pressure response rate | Up to 6 weeks after start of treatment
Change from baseline in pulse pressure | Pre-dose, up to 6 weeks after start of treatment
Number of patients with adverse events | Up to 6 weeks